CLINICAL TRIAL: NCT01570387
Title: A Phase I/II Trial of Pomalidomide and Dexamethasone in Subjects With Previously-Treated AL Amyloidosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-31082; PO-AMYL-PI-0024 (Other: Celgene Corporation)
Record Dates: First submitted 2012-02-27; First posted 2012-04-04 (Estimated); Results first posted 2019-12-16 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: AL Amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — pomalidomide; Dexamethasone; dexamethasone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase I - cohort 1 (Pomalidomide 2mg) plus Dexamethasone (Experimental): Pomalidomide 2 mg/day on days 1-28 plus dexamethasone 10-20 mg on days 1-21 of a 28 day cycle
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone
- Phase I - cohort 2 (Pomalidomide 3mg) plus Dexamethasone (Experimental): Pomalidomide 3 mg/day on days 1-28 plus dexamethasone 10-20 mg on days 1-21 of a 28 day cycle
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone
- Phase I - cohort 3 (Pomalidomide 4mg) plus Dexamethasone (Experimental): Pomalidomide 4 mg/day on days 1-28 plus dexamethasone 10-20 mg on days 1-21 of a 28 day cycle
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone
- Phase II Expansion- (Pomalidomide 4mg) plus Dexamethasone (Experimental): Expansion Phase:
  Pomalidomide 4 mg/day on days 1-28 plus dexamethasone 10-20 mg on days 1-21 of a 28 day cycle
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Pomalidomide — Cohort 1 = 2 mg/day, Cohort 2 = 3 mg/day, Cohort 3 = 4 mg/day: Days 1-21 of a 28 day cycle
  Other Names: pomalyst; imnovist
Drug: Dexamethasone — 10-20 mg on days 1, 8, 15, and 22
  Other Names: Dexamethasone Acetate

SUMMARY:
This study seeks to enroll patients with AL amyloidosis, for whom treatment with one of the standard melphalan chemotherapy-based regimens is either not recommended or is not their preference.

Pomalidomide (CC-4047) is a drug given by mouth, which can change or regulate the functioning of the immune system. So, in theory, it may reduce or prevent the production of the amyloid protein. Pomalidomide is not currently FDA-approved for AL Amyloidosis. Pomalidomide is chemically similar to thalidomide and lenalidomide, both of these drugs have been approved by the FDA for treatment of patients with multiple myeloma (MM), a disease similar to AL Amyloidosis.

Participants in this study will receive pomalidomide and dexamethasone. Phase I is a dose-escalation study and dose escalation will proceed through 3 dose-levels according to standard rules in which dose levels are started sequentially after complete evaluation of the occurrence of dose-limiting toxicities. In the Phase II portion, participants will receive pomalidomide and dexamethasone using the defined maximum tolerated dose.

DETAILED DESCRIPTION:
Primary objective:

Determine dose-limiting toxicity (DLT) and the maximal tolerated dose (MTD) of pomalidomide combined with dexamethasone in subjects with previously- treated light-chain (AL)-amyloidosis

Secondary objectives:

Determine the following at the MTD:

* Hematological complete (CR) very good partial (VGPR) and partial (PR) rates
* duration of response
* organ response
* Time-to-event
* Survival

Exploratory study objective:

To investigate the relationship of changes in the levels of the biomarkers B-type natriuretic peptide (BNP) and troponin I to frequency of specific adverse events and the occurrence of DLT

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign informed consent form.
2. ≥18yrs old
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Biopsy proven tissue amyloid deposits or positive fat aspirate
5. Proof of AL type (a or b)
6. Measurable plasma cell dyscrasia (a or b and c of the following required):

   1. Monoclonal protein in the serum or urine by immunofixation electrophoresis
   2. Plasmacytosis of bone marrow (<30% plasma cells) with monoclonal staining for kappa or lambda light-chain isotype
   3. dFLC of 50mg/L (dFLC=difference in involved and uninvolved serum free light-chain levels)
7. Must have received ≥1 prior treatment for AL amyloidosis, if it is intensive chemotherapy and an autotransplant it must be ≥6 months prior to enrollment on this study
8. Must have recovered from the reversible side effects of any prior therapy; permanent and stable side effects/changes are acceptable. Prior treatment for AL amyloidosis with chemotherapy, thalidomide, lenalidomide or steroids is not an exclusion
9. Eastern Cooperative Group (ECOG) performance status ≤2 at study entry
10. Lab test results within these ranges:

    d. Neutrophil ≥1.5 x10e9/L e. Platelets ≥100x10e9/L f. Total bilirubin <1.5mg/dL g. Aspartate aminotransferase (AST or SGOT) and Alanine Aminotransferase (ALT or SGPT) < 2 x Upper limit of normal h. Serum creatinine <2.5mg/dL
11. Disease free of prior malignancies for at least 5yrs with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in-situ" of the cervix or breast.
12. Females of childbearing potential (FCBP) (a FCBP is a sexually mature woman who has not undergone a hysterectomy or bilateral oophorectomy, or has not been naturally postmenopausal for at least 24 consecutive months) must have a negative serum or urine pregnancy test with a sensitivity ≥ 50 milli-International unit/mL 10-14 days prior to and again ≤ 24 hours of starting pomalidomide and must either commit to continued abstinence from heterosexual intercourse or begin two (2) acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, ≥ 28 days before she starts taking pomalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a vasectomy. All subjects must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
13. Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (subjects intolerant to aspirin may use warfarin or low molecular weight heparin).

Exclusion Criteria:

1. Secondary or familial amyloidosis
2. Multiple myeloma (≥30% plasma cells in a bone marrow biopsy specimen or lytic bone lesions)
3. Cytotoxic chemo or radiation therapy ≤4 weeks of study entry or following baseline evaluation
4. Symptomatic cardiac arrhythmias or O2-dependent restrictive cardiomyopathy
5. Dialysis-dependent
6. Untreated or uncontrolled infections.
7. Serious medical conditions, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
8. Pregnant or breast feeding females (lactating females must agree not to breast feed while taking pomalidomide).
9. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
10. Use of any other experimental drug or therapy within 28 days of baseline.
11. Known intolerance to steroids.
12. Known hypersensitivity to thalidomide or lenalidomide
13. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
14. Concurrent use of other anti-cancer agents or treatments.
15. Known HIV positivity is not an exclusion, unless cluster of differentiation 4 (CD4) counts <200/microliter and/or patient has multi-drug resistant HIV infections and/or other concurrent AIDS-defining conditions. HIV b-DNA < 75 copies/mL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vaishali Sanchorawala, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanchorawala V, Shelton AC, Lo S, Varga C, Sloan JM, Seldin DC. Pomalidomide and dexamethasone in the treatment of AL amyloidosis: results of a phase 1 and 2 trial. Blood. 2016 Aug 25;128(8):1059-62. doi: 10.1182/blood-2016-04-710822. Epub 2016 Jul 5. PMID 27381904

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol was open to accrual between January 2012 and August 2016. Participants were recruited from within the amyloidosis clinic within Boston Medical Center.
Groups:
- Experimental: Phase I - Cohort 1 (Pomalidomide 2mg): Drug: Pomalidomide Cohort 1 = 2 mg/day, Days 1-28
  Drug: Dexamethasone 10-20 mg on days 1, 8, 15, and 22
- Experimental: Phase I - Cohort 2 (Pomalidomide 3mg): Drug: Pomalidomide Cohort 12= 3 mg/day, Days 1-28
  Drug: Dexamethasone 10-20 mg on days 1, 8, 15, and 22
- Experimental: Phase I - Cohort 3 (Pomalidomide 4mg): Drug: Pomalidomide Cohort 3 = 4 mg/day, Days 1-28
  Drug: Dexamethasone 10-20 mg on days 1, 8, 15, and 22
- Experimental: Phase II Expansion- Maximum Tolerated Dose: Drug: Pomalidomide Expansion Phase - Maximum Tolerated Dose = 4 mg/day, Days 1-28
  Drug: Dexamethasone 10-20 mg on days 1, 8, 15, and 22
Period: Overall Study
Arm/Group | Experimental: Phase I - Cohort 1 (Pomalidomide 2mg) | Experimental: Phase I - Cohort 2 (Pomalidomide 3mg) | Experimental: Phase I - Cohort 3 (Pomalidomide 4mg) | Experimental: Phase II Expansion- Maximum Tolerated Dose
Started | 6 | 3 | 6 | 12
Dose Limiting Toxicity | 0 | 0 | 6 | 12
Response to Maximal Tolerated Dose | 0 | 0 | 3 | 6
Completed | 5 | 3 | 6 | 10
Not Completed | 1 | 0 | 0 | 2
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Number of participants in each arm
Groups:
- Phase I - Cohort 1 (Pomalidomide 2mg) Plus Dexam: Pomalidomide: Cohort 1 = 2 mg/day, Cohort 2 = 3 mg/day, Cohort 3 = 4 mg/day: Days 1-28
  Dexamethasone: 10-20 mg on days 1, 8, 15, and 22
- Phase I - Cohort 2 (Pomalidomide 3mg): Pomalidomide 3 mg/day on days 1-28 plus dexamethasone 10-20 mg on days 1-21 of a 28 day cycle
- Phase I - Cohort 3 (Pomalidomide 4mg): Pomalidomide 4 mg/day on days 1-28 plus dexamethasone 10-20 mg on days 1-21 of a 28 day cycle
- Phase II Expansion- (Pomalidomide 4mg) Plus Dexa: Pomalidomide 4 mg/day (MTD) on days 1-28 plus dexamethasone 10-20 mg on days 1-21 of a 28 day cycle
- Total: Total of all reporting groups
Arm/Group | Phase I - Cohort 1 (Pomalidomide 2mg) Plus Dexam | Phase I - Cohort 2 (Pomalidomide 3mg) | Phase I - Cohort 3 (Pomalidomide 4mg) | Phase II Expansion- (Pomalidomide 4mg) Plus Dexa | Total
Number analyzed (Participants) | 6 | 3 | 6 | 12 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 0 | 1 | 5 | 9
  >=65 years | 3 | 3 | 5 | 7 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 1 | 5 | 11
  Male | 2 | 2 | 5 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 3 | 6 | 11 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 6 | 2 | 5 | 11 | 24
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Prior treatments [Count of Participants; unit: Participants] — Number of treatment regimens patients had prior to study enrollment
  Participants
    1 to 2 prior treatments | 4 | 3 | 1 | 8 | 16
    greater than 2 prior treatments | 2 | 0 | 5 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Assessing Dose-limiting Toxicity to Determine Maximal Tolerated Dosage at 2 Milligram Dose
Description: Number of patients in Phase I cohort 1 experiencing dose-limiting toxicity at the 2 milligram dose of pomalidomide combined with dexamethasone in subjects with previously- treated light-chain amyloidosis
Time Frame: one month
Measure: Count of Participants; unit: Participants
Groups:
- Pom Plus Dex: Pomalidomide dexamethasone
  Pomalidomide: Cohort 1 = 2 mg/day, Cohort 2 = 3 mg/day, Cohort 3 = 4 mg/day: Days 1-28
  Dexamethasone: 10-20 mg on days 1, 8, 15, and 22
Arm/Group | Pom Plus Dex
Number analyzed (Participants) | 6
Participants | 0

2. Primary Outcome: Assessing Dose-limiting Toxicity to Determine Maximal Tolerated Dosage at 3 Milligram Dose
Description: Number of patients in Phase I cohort 2 experiencing dose limiting toxicity in the 3 milligram dose level, cohort 2.
Time Frame: One month
Measure: Count of Participants; unit: Participants
Arm/Group | Pom Plus Dex
Number analyzed (Participants) | 3
Participants | 0

3. Primary Outcome: Assessing Dose-limiting Toxicity to Determine Maximal Tolerated Dosage at 4 Milligram Dose
Description: Number of patients in Phase I cohort 3 experiencing dose-limiting toxicity at the 4 milligram dose for participants within the third dose cohort
Time Frame: One month
Measure: Count of Participants; unit: Participants
Arm/Group | Pom Plus Dex
Number analyzed (Participants) | 6
Participants | 1

4. Secondary Outcome: Response to the Maximal Tolerated Dose
Description: Number of participants with a response to treatment at that maximal tolerated dose (including partial, very good, or complete responses)
Time Frame: one year
Population: Number of evaluable patients treated at the maximal tolerated dose of 4mg including the Phase I cohort 3 participants and the Phase II expansion participants
Measure: Count of Participants; unit: Participants
Arm/Group | Pom Plus Dex
Number analyzed (Participants) | 18
Participants | 10

ADVERSE EVENTS:
Time Frame: 6 years
Description: Adverse events for each participant were assessed at all visits while treatment continued through 30 days post last dose. 6 years represents the time from first participant initiating treatment though last participant completing treatment.
Groups:
- Phase I - Cohort 1 (Pomalidomide 2mg): Drug: Pomalidomide Cohort 1 = 2 mg/day, Days 1-28
  Drug: Dexamethasone 10-20 mg on days 1, 8, 15, and 22
- Phase I - Cohort 2 (Pomalidomide 3mg): Drug: Pomalidomide Cohort 2 = 3 mg/day, Days 1-28
  Drug: Dexamethasone 10-20 mg on days 1, 8, 15, and 22
- Phase I - Cohort 3 (Pomalidomide 4mg): Drug: Pomalidomide Cohort 3 = 4 mg/day, Days 1-28
  Drug: Dexamethasone 10-20 mg on days 1, 8, 15, and 22
- Phase II Expansion- Maximum Tolerated Dose: Drug: Pomalidomide Maximum Tolerated Dose = 4 mg/day, Days 1-28
  Drug: Dexamethasone 10-20 mg on days 1, 8, 15, and 22
Arm/Group | Phase I - Cohort 1 (Pomalidomide 2mg) | Phase I - Cohort 2 (Pomalidomide 3mg) | Phase I - Cohort 3 (Pomalidomide 4mg) | Phase II Expansion- Maximum Tolerated Dose
All-Cause Mortality (participants affected / at risk) | 1/6 | 0/3 | 0/6 | 1/12
Serious Adverse Events (participants affected / at risk) | 2/6 | 0/3 | 3/6 | 3/12
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 6/6 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I - Cohort 1 (Pomalidomide 2mg) (N=6) | Phase I - Cohort 2 (Pomalidomide 3mg) (N=3) | Phase I - Cohort 3 (Pomalidomide 4mg) (N=6) | Phase II Expansion- Maximum Tolerated Dose (N=12)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
sepsis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I - Cohort 1 (Pomalidomide 2mg) (N=6) | Phase I - Cohort 2 (Pomalidomide 3mg) (N=3) | Phase I - Cohort 3 (Pomalidomide 4mg) (N=6) | Phase II Expansion- Maximum Tolerated Dose (N=12)
White blood cell count decreased (Investigations) | 3 (3) | 0 (0) | 1 (4) | 10 (15)
wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
weakness (General disorders) | 3 (3) | 1 (1) | 3 (4) | 4 (5)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
visual blurring (Eye disorders) | 4 (4) | 0 (0) | 1 (1) | 3 (3)
urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
urinary incontinence (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
urinary frequency (Renal and urinary disorders) | 4 (5) | 0 (0) | 4 (5) | 0 (0)
urinary hesitancy (Renal and urinary disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (2)
hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (12) | 5 (6)
upper respiratory infection (Infections and infestations) | 2 (3) | 1 (2) | 4 (6) | 3 (4)
hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (4) | 2 (2)
tremor (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 4 (5)
tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
platelet count decreased (Investigations) | 2 (5) | 0 (0) | 2 (2) | 4 (9)
sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 5 (7)
pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
paresthesia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (2) | 2 (3)
palpitations (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 5 (6)
pain-extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2)
arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 6 (9) | 9 (16)
nausea (Gastrointestinal disorders) | 2 (2) | 2 (3) | 3 (5) | 4 (4)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
muscle disorder - cramping (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 4 (4) | 3 (3)
mood alteration (Psychiatric disorders) | 3 (3) | 0 (0) | 2 (2) | 2 (2)
lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 5 (18) | 5 (9)
lightheadedness (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
leukocyte count decreased (Investigations) | 0 (0) | 1 (1) | 4 (5) | 1 (1)
insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 4 (5)
infection - skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (4) | 3 (9)
hyponatremia (Metabolism and nutrition disorders) | 3 (9) | 0 (0) | 2 (2) | 4 (4)
hypoalbuminemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 5 (7) | 2 (3)
hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
hyperkalemia (Metabolism and nutrition disorders) | 3 (6) | 0 (0) | 3 (4) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 6 (12) | 2 (4)
hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 2 (3) | 4 (4)
fever (General disorders) | 1 (1) | 0 (0) | 5 (5) | 2 (2)
fatigue (General disorders) | 3 (4) | 2 (2) | 4 (8) | 8 (10)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
edema - limbs (General disorders) | 0 (0) | 0 (0) | 2 (2) | 7 (9)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 5 (10) | 6 (6)
dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 2 (3) | 0 (0)
dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 2 (3) | 2 (4)
diarrhea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 3 (5) | 3 (4)
creatinine elevated (Investigations) | 4 (8) | 1 (1) | 5 (8) | 5 (10)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (4) | 4 (6)
constipation (Gastrointestinal disorders) | 4 (5) | 3 (3) | 3 (3) | 4 (4)
chronic kidney disease (Renal and urinary disorders) | 2 (4) | 0 (0) | 2 (5) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 3 (5)
anemia (Investigations) | 5 (8) | 1 (2) | 4 (15) | 6 (8)
anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 2 (2) | 3 (5)
abdominal bloating (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
hypokalemia (Investigations) | 1 (2) | 0 (0) | 2 (2) | 0 (0)
hematuria (Renal and urinary disorders) | 0 (0) | 1 (2) | 2 (2) | 0 (0)
heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
hemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
chest pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
chills (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
aspartate aminotransferase increased (Investigations) | 5 (5) | 0 (0) | 2 (2) | 4 (4)
anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-11): https://cdn.clinicaltrials.gov/large-docs/87/NCT01570387/Prot_SAP_000.pdf